CLINICAL TRIAL: NCT01950117
Title: Complete Removal of Neoplastic Large Colorectal Polyps: a Prospective Randomized Comparison of Endoscopic Mucosal Resection or Conventional Polypectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Showa Inan General Hospital (Other)
Responsible Party: Principal Investigator, Akira Horiuchi, Chief, Digestive Disease Center, Showa Inan General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMR vs. polypectomy
Record Dates: First submitted 2013-09-21; First posted 2013-09-25 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Colorectal Polyps
Keywords: nonpedunculated; neoplastic; colorectal; polyps
MeSH Terms: conditions — Polyps | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional polypectomy (Active Comparator): Colorectal polyps from 10 mm to 25 mm was found. Submucosal injection of saline solution before removal was not performed for polypectomy. The snare used for polypectomy was a dual loop wire snare with a loop size of 33/16 mm (SN-3316LX, Medico's Hirata Inc., Osaka, Japan). An ERBE ICC200 (Amco, Tokyo, Japan) was used in the Endocut mode with the effect 3 current set at output limit 120W and forced coagulation current set at output limit 35W for conventional polypectomy. Prophylactic clipping after polyp removal was routinely performed.
  Interventions: Procedure: Conventional polypectomy
- Endoscopic mucosal resection (Experimental): Colorectal polyp from 10 mm to 25 mm was found. Submucosal injection of saline solution before removal was performed for EMR. The snare used for EMR was a dual loop wire snare with a loop size of 33/16 mm (SN-3316LX, Medico's Hirata Inc., Osaka, Japan). An ERBE ICC200 (Amco, Tokyo, Japan) was used in the Endocut mode with the effect 3 current set at output limit 120W and forced coagulation current set at output limit 35W for EMR. Prophylactic clipping after polyp removal was routinely performed.
  Interventions: Procedure: Endoscopic mucosal resection

INTERVENTIONS:
Procedure: Endoscopic mucosal resection — Nonpedunculated neoplastic colorectal polyps from 10 mm to 25 mm in diameter were resected after submucosal injection of saline solution before removal.
  Arms: Endoscopic mucosal resection
Procedure: Conventional polypectomy — Nonpedunculated neoplastic colorectal polyps from 10 mm to 25 mm in diameter were resected using conventional polypectomy. Submucosal injection of saline solution before removal was not performed.
  Arms: Conventional polypectomy

SUMMARY:
Recently, it was reported that the incomplete resection rate of neoplastic large polyps after conventional polypectomy was markedly high in clinical practice. The incomplete resection rate of neoplastic large polyps after endoscopic mucosal resection (EMR) is not known.

The aim of this study is to compare the incomplete resection rate of neoplastic large polyps after EMR or conventional polypectomy. The EMR technique is preferable to conventional polypectomy for the complete resection of the large polyps (>15 mm in diameter)

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were nonpedunculated neoplastic colorectal polyps from 10 mm to 25 mm in diameter.

Exclusion Criteria:

* less than 20 years old, history of previous colorectal surgical resection, American Society of Anesthesiologists class III and IV, allergic to propofol used or its components (soybeans or eggs), or poor bowel preparation.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The incomplete resection rate of neoplastic polyps as determined by the histopathologic examination. | Two weeks

SECONDARY OUTCOMES:
Postpolypectomy bleeding requiring endoscopic intervention within two weeks after polypectomy | Two weeks

OTHER OUTCOMES:
the procedure time | One day

CONTACTS AND LOCATIONS:
Locations (1):
- Showa Inan General Hospital, Komagane, Nagano, Japan